CLINICAL TRIAL: NCT02459418
Title: Comparative Pharmacokinetics of AFOLIA and US Gonal-f® RFF Redi-ject After Single Subcutaneous Application. A Randomised, Open Label, 2-way Cross-over Study
Brief Title: Comparative Pharmacokinetics of AFOLIA and US Gonal-f® RFF Redi-ject After Single Subcutaneous Application
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fertility Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FIN1002
Record Dates: First submitted 2015-05-19; First posted 2015-06-02 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Healthy Volunteers
Keywords: Afolia; Follitropin
MeSH Terms: interventions — follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Afolia - US Gonal-f® (Sequence A) Arm (Experimental): During the Cross-Over Pharmacokinetic Phase, subjects will be randomly assigned to receive treatment sequence: (Sequence A): Single subcutaneous injection of 225IU Afolia on study day 1, followed by a single subcutaneous injection of 225IU US Gonal-f® on study day 27.
  Interventions: Drug: Afolia; Drug: US Gonal-f®
- US Gonal-f® - Afolia (Sequence B) Arm: (Active Comparator): During the Cross-Over Pharmacokinetic Phase, patients will be randomly assigned to receive treatment sequence (Sequence B): Single subcutaneous injection of 225IU US Gonal-f® on study day 1, followed by a single subcutaneous injection of 225IU Afolia on study day 27
  Interventions: Drug: Afolia; Drug: US Gonal-f®

INTERVENTIONS:
Drug: Afolia — During the Cross-Over Pharmacokinetic Phase, subjects will be randomly assigned to receive one of the following treatment sequences:
  Sequence A: Single subcutaneous injection of 225IU Afolia on study day 1, followed by a single subcutaneous injection of 225IU US Gonal-f® on study day 27.
  Sequence B: Single subcutaneous injection of 225IU US Gonal-f® on study day 1, followed by a single subcutaneous injection of 225IU Afolia on study day 27
  Other Names: Follitropin Alfa
Drug: US Gonal-f® — During the Cross-Over Pharmacokinetic Phase, subjects will be randomly assigned to receive one of the following treatment sequences:
  Sequence A: Single subcutaneous injection of 225IU Afolia on study day 1, followed by a single subcutaneous injection of 225IU US Gonal-f® on study day 27.
  Sequence B: Single subcutaneous injection of 225IU US Gonal-f® on study day 1, followed by a single subcutaneous injection of 225IU Afolia on study day 27
  Other Names: Follitropin Alfa

SUMMARY:
Comparative PK study after single SC application of Afolia and the reference product (US Gonal-f®). Objective: To demonstrate equivalence within 80%-125% margin of the reference product for the area under the curve (AUC) of Afolia.

DETAILED DESCRIPTION:
To demonstrate equivalence within the 80% to 125% margin of the reference product for the baseline corrected area under the follicle-stimulating hormone (FSH) serum concentration-time curve from time zero to the last quantifiable concentration of AFOLIA compared to the reference product (United States [US] Gonal-f® RFF)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female volunteers aged 18 to 42 years (inclusive) with a Body mass index of 18.0 to 32.0 kg/m2 (inclusive)
2. Subjects who have used oral contraceptives for at least 3 months before study entry and are prepared to stop taking oral contraception from screening and to use effective non-hormonal methods of birth control until completion of 1 menstrual cycle after the last dose administration
3. Women of child bearing potential must agree to use effective non-hormonal contraception for birth control until completion of 1 menstrual cycle after the last dose administration
4. Subjects with a regular menstruation cycle (25 to 34 days) before initiation of oral contraception
5. Subjects with both ovaries
6. Subjects who are negative for drugs of abuse and alcohol tests at screening and each admission
7. Subjects who are healthy as determined by pre study medical history, physical examination and 12-Lead electrocardiogram (ECG)
8. Subjects whose clinical laboratory test results are not clinically relevant and are acceptable to the investigator
9. Subjects who are able and willing to give written informed consent

Exclusion Criteria:

1. Subjects who do not conform to the above inclusion criteria
2. Subjects with polycystic ovary syndrome
3. Subjects with developing follicles or solid ovarian cysts >2 cm or complex cysts regardless of size
4. Subjects with a history of hypersensitivity to FSH (Ovary Hyperstimulation Syndrome)
5. Subjects with impaired thyroid function (treated or untreated)
6. Subjects with a history of malignant disease
7. Subjects with aspartate aminotransferase and/or alanine aminotransferase >2 x upper limit of normal reference range
8. Subjects with other clinically relevant findings (ECG, blood pressure, physical, laboratory examination)
9. Subjects with a smoking history of more than 5 cigarettes per day
10. Subjects with evidence of abuse of drugs or alcoholic beverages
11. Subjects with a positive screen for hepatitis B surface antigen, antibodies to the hepatitis C virus or antibodies to the human immunodeficiency virus 1/2
12. Subjects who have participated in a clinical trial within the 3 months prior to this study
13. Subjects who are unlikely to co-operate with the requirements of the study
14. Subjects with symptoms of a clinically relevant illness during the 3 weeks prior to study day -1
15. Subjects who are pregnant, lactating or attempting to become pregnant
16. Subjects with any medical condition (including a known predisposition to porphyria) that, in the opinion of the investigator, could interfere with safety of the subject or interfere with the objectives of the study
17. Subjects who are vegans or have medical dietary restrictions
18. Subjects who cannot communicate reliably with the investigator

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Jenkins, DM FRCOG, Study Director — Fertility Biotech AG
Locations (1):
- Quintiles Drug Research Unit at Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 1, randomised, open label, 2-period, 2-treatment, crossover study in healthy female subjects. 42 subjects were randomised to receive either AFOLIA on study day 1 and Gonal-f® RFF on study day 27 or Gonal-f® RFF on study day 1 and AFOLIA on study day 27.
Pre-assignment Details: Screening was conducted at more than 1 visit to the clinical unit during study days -28 to -1 to allow completion of all assessments. Only subjects taking oral contraception for at least 3 months could enter the study. Subjects were required to stop taking their regular oral contraceptives so they could receive LupronDepot®.
Groups:
- AFOLIA Then Gonal-f® RFF: On study day -1 (10 days after administration of LupronDepot®) subjects were assessed for eligibility of treatment by confirmation of down regulation of endogenous FSH levels. If down regulation was not confirmed the evaluation may have been repeated up to 7 days later.
  Period 1: On study day 1, eligible subjects received a single subcutaneous (s.c.) dose of the first FSH preparation, 225 International Units (IU) AFOLIA, in the abdomen. On study day 16, subjects received a second LupronDepot® intramuscular (i.m.) injection.
  Period 2: On study day 26, subjects underwent a further FSH down regulation assessment. This evaluation was repeated up to 7 days later if required and if down regulation was not confirmed after the second evaluation, the subject was no longer able to continue in the study. If eligibility was confirmed, the subject received the alternative FSH preparation, 225 IU Gonal-f® RFF, on study day 27. Exit examinations were performed on study day 35.
- Gonal-f® RFF Then AFOLIA: On study day -1 (10 days after administration of LupronDepot®) subjects were assessed for eligibility of treatment by confirmation of down regulation of endogenous FSH levels. If down regulation was not confirmed the evaluation may have been repeated up to 7 days later.
  Period 1: On study day 1, eligible subjects received a single s.c. dose of the first FSH preparation, 225 IU Gonal-f® RFF, in the abdomen. On study day 16, subjects received a second LupronDepot® i.m. injection.
  Period 2: On study day 26, subjects underwent a further FSH down regulation assessment. This evaluation was repeated up to 7 days later if required and if down regulation was not confirmed after the second evaluation, the subject was no longer able to continue in the study. If eligibility was confirmed, the subject received the alternative FSH preparation of 225 IU AFOLIA on study day 27. Exit examinations were performed on study day 35.
Period: Overall Study
Arm/Group | AFOLIA Then Gonal-f® RFF | Gonal-f® RFF Then AFOLIA
Started | 21 | 21
Received First Treatment | 21 | 21
Received Second Treatment | 13 | 15
Completed | 13 | 15
Not Completed | 8 | 6
Not completed — Exclusion Criteria | 4 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Endometrial thickness of >5 mm | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Elevated Creatine Kinase | 1 | 0
Not completed — Abnormal Transvaginal Ultrasound | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects randomized to receive study treatment.
Groups:
- AFOLIA Then Gonal-f® RFF: On study day -1 (10 days after administration of LupronDepot®) subjects were assessed for eligibility of treatment by confirmation of down regulation of endogenous FSH levels. If down regulation was not confirmed the evaluation may have been repeated up to 7 days later.
  Period 1: On study day 1, eligible subjects received a single s.c. dose of the first FSH preparation, 225 International Units (IU) AFOLIA, in the abdomen. On study day 16, subjects received a second LupronDepot® i.m. injection.
  Period 2: On study day 26, subjects underwent a further FSH down regulation assessment. This evaluation was repeated up to 7 days later if required and if down regulation was not confirmed after the second evaluation, the subject was no longer able to continue in the study. If eligibility was confirmed, the subject received the alternative FSH preparation, 225 IU Gonal-f® RFF on study day 27.
  Exit examinations were performed on study day 35.
- Total: Total of all reporting groups
Arm/Group | AFOLIA Then Gonal-f® RFF | Gonal-f® RFF Then AFOLIA | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 27.8 [18 to 39] | 28.1 [18 to 37] | 28.0 [18 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Baseline Corrected FSH Area Under the Serum Concentration-time Curve From Zero to the Last Quantifiable Measurement [AUC(0-last)]
Description: AUC(0-last) was estimated for baseline corrected FSH in serum by noncompartmental methods using actual elapsed time from dosing. Baseline corrected concentrations were determined by subtracting the baseline concentration (collected immediately prior to dosing in that period) from the postdose concentration.
  Geometric mean baseline corrected FSH exposure results are presented for all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PK time point after administration of AFOLIA or Gonal-f® RFF.
Time Frame: From 0 (predose),0.5, 1, 3, 6, 9, 12, 16, 20, 21, 22, 23, 24, 25, 26, 27, 28, 48, 72, 96, 120, 144, 168 and 192 hours postdose.
Population: Analysis was performed on the Pharmacokinetic Analysis Set (PKAS) which includes all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PK time point after administration of AFOLIA or Gonal-f® RFF. Only subjects with concentration data for determination of AUC(0-last) are included.
Measure: Geometric Mean (Full Range); unit: nanograms*hours/mL (ng*h/mL)
Groups:
- AFOLIA: All subjects who received the test product 225 IU AFOLIA and had at least 1 measured concentration at a scheduled pharmacokinetic (PK) or pharmacodynamic (PD) time point after administration of AFOLIA.
- Gonal-f® RFF: All subjects who received the test product 225 IU Gonal-f® RFF and had at least 1 measured concentration at a scheduled PK or PD time point after administration of Gonal-f® RFF.
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 36 | 33
nanograms*hours/mL (ng*h/mL) | 18.96 [2.2 to 73.2] | 10.47 [0.288 to 42.8]
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; A mixed-effects analysis of variance (ANOVA) model with sequence, treatment and period as fixed effects, and subject nested within sequence as random effect was used. Least squares (LS) means and 90% confidence intervals (CIs) for treatment differences on log-scale were obtained and back transformed to provide geometric LS mean ratios of AFOLIA over Gonal-f® RFF; Test type: Equivalence — The 90% CIs of the ratios of geometric means of log-transformed baseline corrected AUC(0-last) were used to assess bioequivalence between Gonal-f® RFF and AFOLIA using the bioequivalence interval of 80.00% to 125.00%; Geometric LS Mean Ratio = 164.96, 90% CI 2-sided [137.82 to 197.45]

2. Primary Outcome: Baseline Corrected FSH Maximum Serum Concentration (Cmax)
Description: Cmax was estimated for baseline corrected FSH in serum by noncompartmental methods using actual elapsed time from dosing. Baseline corrected concentrations were determined by subtracting the baseline concentration (collected immediately prior to dosing in that period) from the postdose concentration.
  Geometric mean baseline corrected FSH exposure results are presented for all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PK time point after administration of AFOLIA or Gonal-f® RFF.
Time Frame: From 0 hours (predose) to 192 hours postdose.
Population: This analysis was performed on the PKAS which includes all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PK time point after administration of AFOLIA or Gonal-f® RFF. Only subjects with concentration data for determination of Cmax are included.
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- AFOLIA: All subjects who received the test product AFOLIA and had at least 1 measured concentration at a scheduled PK or PD time point after administration of AFOLIA.
- Gonal-f® RFF: All subjects who received the test product Gonal-f® RFF and had at least 1 measured concentration at a scheduled PK or PD time point after administration of Gonal-f® RFF.
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 36 | 34
ng/mL | 0.4795 [0.21 to 1.13] | 0.3692 [0.048 to 1.17]
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; An ANOVA model with sequence, treatment and period as fixed effects, and subject nested within sequence as random effect was used. LS means and 90% CIs for treatment differences on log-scale were obtained and back-transformed to provide geometric LS mean ratios of AFOLIA over Gonal-f® RFF; Test type: Equivalence — The 90% CIs of the ratios of geometric means of log-transformed baseline corrected Cmax were used to assess bioequivalence between Gonal-f® RFF and AFOLIA using the bioequivalence interval of 80.00% to 125.00%; Geometric LS Mean Ratio = 123.15, 90% CI 2-sided [108.12 to 140.28]

3. Secondary Outcome: Baseline Corrected FSH Area Under the Serum Concentration-time Curve Extrapolated to Infinity [AUC(0-∞)]
Description: AUC(0-∞) was estimated for baseline corrected FSH in serum by noncompartmental methods using actual elapsed time from dosing. Baseline corrected concentrations were determined by subtracting the baseline concentration (collected immediately prior to dosing in that period) from the postdose concentration.
  Geometric mean baseline corrected FSH exposure results are presented for all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PK time point after administration of AFOLIA or Gonal-f® RFF.
Time Frame: From 0 hours (predose) to 192 hours postdose.
Population: This analysis was performed on the PKAS which includes all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PK time point after administration of AFOLIA or Gonal-f® RFF. Only subjects with suitable terminal phase profiles for determination of AUC(0-∞) are included.
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Groups:
- AFOLIA: All subjects who received the test product 225 IU AFOLIA and had at least 1 measured concentration at a scheduled PK or PD time point after administration of AFOLIA.
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 18 | 12
ng*h/mL | 27.88 [10.8 to 76] | 20.57 [6.43 to 49]
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — The 90% CIs of the ratios of geometric means of log-transformed baseline corrected AUC(0-∞) were used to assess bioequivalence between Gonal-f® RFF and AFOLIA using the bioequivalence interval of 80.00% to 125.00%; Geometric LS mean ratio = 133.68, 90% CI 2-sided [102.42 to 174.49]

4. Secondary Outcome: Baseline Corrected Time to Reach Maximum FSH Serum Concentration (Tmax)
Description: Tmax was estimated for baseline corrected FSH in serum by noncompartmental methods using actual elapsed time from dosing. Baseline corrected concentrations were determined by subtracting the baseline concentration (collected immediately prior to dosing in that period) from the postdose concentration.
  Geometric mean was not calculated for Tmax and the non-transformed results are presented are for all subjects who received active study drug and had Tmax estimated in both periods.
Time Frame: From 0 hours (predose) to 192 hours postdose.
Population: This analysis was performed on the PKAS which includes all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PK time point after administration of AFOLIA or Gonal-f® RFF. Only subjects with Tmax estimated in both periods are included.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 36 | 34
hours | 24.05 [6 to 28.03] | 16 [3 to 28.08]
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; Non-transformed Tmax was tested using the non-parametric Wilcoxon signed rank test to assess the differences between Gonal-f® RFF and AFOLIA. Median differences and corresponding 90% CIs were calculated using an exact Hodges-Lehmann estimate; Test type: Other; Median Difference (Net) = 7.5, 90% CI 2-sided [4.5 to 11.5]

5. Secondary Outcome: Baseline Corrected FSH Apparent Terminal Half-life
Description: Apparent terminal half-life was defined as ln2/apparent terminal rate constant (λz). λz is determined by linear regression of the terminal points of the log-linear concentration-time curve. Visual assessment was used to identify the terminal linear phase of the baseline corrected concentration-time profile. A minimum of 3 data points was used for determination.
  Terminal half-life was estimated for baseline corrected FSH in serum by noncompartmental methods using actual elapsed time from dosing. Baseline corrected concentrations were determined by subtracting the baseline concentration (collected immediately prior to dosing in that period) from the postdose concentration.
  Geometric mean baseline corrected FSH exposure results are presented for all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PK time point after administration of AFOLIA or Gonal-f® RFF.
Time Frame: From 0 hours (predose) to 192 hours postdose.
Population: This analysis was performed on the PKAS which includes all subjects who received active study drug and had at least 1 measured concentration at a scheduled PK or PD time point after administration of AFOLIA or Gonal-f® RFF. Only subjects with suitable terminal phase profiles for determination of terminal half-life are included.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 18 | 12
hours | 20.4 [7.76 to 62] | 18.02 [7.37 to 61.4]

6. Secondary Outcome: Baseline Corrected 17ß-Estrodiol (E2) Serum Exposure AUC(0-last)
Description: AUC(0-last) was estimated for baseline corrected E2 in serum by noncompartmental methods using actual elapsed time from dosing. Baseline corrected concentrations were determined by subtracting the baseline concentration (collected immediately prior to dosing in that period) from the postdose concentration.
  Geometric mean baseline corrected E2 exposure results are presented for all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PD time point after administration of AFOLIA or Gonal-f® RFF.
Time Frame: From 0 hours (predose) to 192 hours postdose.
Population: This analysis was performed on the PKAS which includes all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PK time point after administration of AFOLIA or Gonal-f® RFF. Only subjects with concentration data for determination of AUC(0-last) are included.
Measure: Geometric Mean (Full Range); unit: pg*h/mL
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 34 | 31
pg*h/mL | 888 [12.4 to 13800] | 570 [7.6 to 11700]
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Mean Ratio = 163, 90% CI 2-sided [94 to 282.67]

7. Secondary Outcome: Baseline Corrected E2 Cmax
Description: Cmax was estimated for baseline corrected E2 in serum by noncompartmental methods using actual elapsed time from dosing. Baseline corrected concentrations were determined by subtracting the baseline concentration (collected immediately prior to dosing in that period) from the postdose concentration.
  Geometric mean baseline corrected E2 exposure results are presented for all subjects who received active study drug and had at least 1 measured and valid concentration at a scheduled PD time point after administration of AFOLIA or Gonal-f® RFF.
Time Frame: From 0 hours (predose) to 192 hours postdose.
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 34 | 34
pg/mL | 28.03 [3.5 to 227.1] | 15.95 [0.1 to 171]
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 177.17, 90% CI 2-sided [125.65 to 249.81]

8. Secondary Outcome: Baseline Corrected E2 Tmax
Description: Tmax was estimated for baseline corrected E2 in serum by noncompartmental methods using actual elapsed time from dosing. Baseline corrected concentrations were determined by subtracting the baseline concentration (collected immediately prior to dosing in that period) from the postdose concentration.
  Geometric mean was not calculated for Tmax and the non-transformed results are presented are for all subjects who received active study drug and had Tmax estimated in both periods.
Time Frame: From 0 hours (predose) to 192 hours postdose.
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | AFOLIA | Gonal-f® RFF
Number analyzed (Participants) | 34 | 34
hours | 47.92 [22 to 96] | 27.5 [20 to 144.5]
Statistical Analysis 1: Comparison: AFOLIA vs Gonal-f® RFF; Non-transformed Tmax was tested using the non-parametric Wilcoxon signed rank test to assess the differences between Gonal-f® RFF and AFOLIA. Median difference and corresponding 90% CIs were was calculated using an Exact Hodges-Lehmann estimate with an exact confidence interval; Test type: Other; Median Difference (Net) = 2.14, 90% CI 2-sided [-9.91 to 12.29]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAEs) were reported from study day 1 to study day 35.
Description: A TEAE was defined as any adverse event that began or worsened following first dose administration. Adverse events (AEs) occurring between treatments were attributed to the last treatment received. Subjects were asked about AEs at each contact with the site (visits and telephone calls).
Groups:
- AFOLIA: This analysis set contained all subjects who received one dose of AFOLIA (225 IU).
- Gonal-f® RFF: This analysis set contained all subjects who received one dose of Gonal-f® RFF (225 IU).
Arm/Group | AFOLIA | Gonal-f® RFF
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 21/36 | 22/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AFOLIA (N=36) | Gonal-f® RFF (N=34)
Hot flush (Vascular disorders) | 11 (11) | 11 (11)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 10 (12)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Catheter site related reaction (General disorders) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contract agreement. Results may not be published or referred to, in whole or in part, without the prior express written consent of the Sponsor.